CLINICAL TRIAL: NCT06609369
Title: Neural Mechanisms Connecting Deficient Sleep and Smoking Relapse
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000037737; R01DA061285 (NIH)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Tobacco Use; Tobacco Cessation; Insomnia
MeSH Terms: conditions — Tobacco Use; Tobacco Use Cessation; Sleep Initiation and Maintenance Disorders | interventions — Varenicline

STUDY DESIGN:
Intervention Model Description: Participants who smoke randomly assigned and stratified by sex and severity of tobacco dependence
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental health intervention (Experimental): Experimental health intervention and varenicline starting 4 weeks before and continuing for 4 weeks after a target quit date for a total of 8 weeks
  Interventions: Behavioral: Experimental health intervention; Drug: Varenicline
- Control health intervention (Active Comparator): Control health intervention and varenicline starting 4 weeks before and continuing for 4 weeks after a target quit date for a total of 8 weeks
  Interventions: Drug: Varenicline

INTERVENTIONS:
Behavioral: Experimental health intervention — Behavioral health intervention
  Arms: Experimental health intervention
Drug: Varenicline — Days 1-3: 0.5mg once daily, Days 4-7: 0.5mg twice daily; Days 8-56: 1.0mg twice daily.

SUMMARY:
The study aims to investigate whether behavioral interventions promote cessation in adult smokers by ameliorating negative emotions and improving self-control and identify the neural markers of these effects.

DETAILED DESCRIPTION:
The primary objectives of this study are to compare the effectiveness of two types of behavioral interventions, when combined with varenicline medication, in promoting tobacco cessation among treatment-seeking adults and to elucidate the underlying mechanisms. The secondary objective of this study is to examine sex differences.

Investigators will recruit from two primary sources: 1) community-based recruitment strategies including web and social media ads, lay community members to recruit, and local communication channels; 2) investigators will invite referred patients to the outpatient Tobacco Treatment Service (TTS) at Yale-New Haven Hospital.

All participants will be assigned to one of two behavioral interventions. Both groups will receive treatment with varenicline and attend weekly individual counseling sessions (standard care or cognitive behavioral therapy for insomnia) and wear research-grade sleep actiwatches for passive sleep monitoring.

Participants will have a total of five expected research visits with a scheduled target quit date for Week 4. Participants will undergo MRI at baseline and at Week 4, and attend follow-ups at week 8, 12, and 26.

ELIGIBILITY:
Inclusion Criteria:

* English literate
* report heavy tobacco use (including nicotine e-cigarettes) for >6 months
* meet biochemical cut off for recent cigarette smoking or e-cigarette use
* optimal body mass index

Exclusion Criteria:

* currently enrolled in other treatments
* neuropsychiatric exclusions that could interfere with study participation, increase risk of adverse events, and/or induce deficient sleep
* medical contraindications for fMRI, varenicline, and/or behavioral treatment
* factors that cause deficient sleep and for which behavioral treatment has less benefit
* women who are pregnant or nursing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Mean number cigarettes smoked per day | Baseline, week 4, 8, 12, and 26
  Mean number cigarettes smoked per day assessed by Time Line Follow Back method
Smoking status | Baseline
  Assess expired breath carbon monoxide (CO) at baseline. CO is a standard biomarker of combustible tobacco use, is sensitive to detecting cigarette substitution, and has a typical half-life of 4 hours, and is a standard biomarker for confirming recent smoking abstinence (CO <5ppm has optimal sensitivity and specificity for biochemically verifying smoking status, including at lower smoking levels).
Quit status | Week 4, 8, 12, and 26
  To inquire whether participants have refrained from tobacco use at each visit following their quit date. The quit status will also be verified by assessing expired breath carbon monoxide (CO). CO is a standard biomarker of combustible tobacco use, is sensitive to detecting cigarette substitution, and has a typical half-life of 4 hours, and is a standard biomarker for confirming recent smoking abstinence (CO <5ppm has optimal sensitivity and specificity for biochemically verifying smoking status, including at lower smoking levels)
Days to smoking relapse | Week 4, 8, 12, and 26
  Days of resuming smoking since Week 4 schedule quit date as assessed by the Time Line Follow-back

SECONDARY OUTCOMES:
Change in PROMIS Sleep Disturbance | Baseline, week 4, 8, 12, and 26
  The PROMIS Sleep Disturbance is an 8 item self-report of perceptions of sleep quality, sleep depth, and restoration associated with sleep. Each item on the measure is rated on a 5-point scale. PROMIS measures are scored on the T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. High scores mean greater severity of sleep disturbance.
Change in PROMIS Sleep-Related Impairment | Baseline, week 4, 8, 12, and 26
  The PROMIS Sleep-Related Impairment is an 8 item self-report of perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness. Each item on the measure is rated on a 4-point scale. The score range is 4 to 32. High scores mean greater severity of sleep related impairment.
Change in Insomnia Severity Index | Baseline, week 4, 8, 12, and 26
  The Insomnia Severity Index is a 7-item brief screening tool for insomnia. Each item on the measure is rated on a 5-point scale (0-4), with a total score range 0-28. High scores mean greater severity of insomnia.

CONTACTS AND LOCATIONS:
Overall Officials: Chiang-Shan Li, Principal Investigator — Yale University; Lisa Fucito, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - Yale University, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No